CLINICAL TRIAL: NCT01905280
Title: Ridge Preservation Comparing the Clinical and Histologic Healing of a PTFE Non-resorbable Membrane Versus an Acellular Dermal Matrix Allograft Plus a Facial Overaly Bovine Xenograft.
Brief Title: Ridge Preservation Comparing 2 Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13.0330
Record Dates: First submitted 2013-07-12; First posted 2013-07-23 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Alveolar Ridge Deficiency
Keywords: allograft; acellular dermal matrix; alveolar ridge
MeSH Terms: interventions — Polytetrafluoroethylene; Alloderm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acellular dermal matrix (Experimental): A ridge preservation graft will be performed and then covered using acellular dermal matrix as a membrane.
  Interventions: Procedure: Acellular dermal matrix
- Non-resorbable membrane (Active Comparator): A ridge preservation graft will be performed and then covered using a non-resorbable PTFE membrane.
  Interventions: Procedure: Non-resorbable membrane

INTERVENTIONS:
Procedure: Non-resorbable membrane — The ridge preservation graft will be covered with a non-resorbable PTFE membrane during the surgery.
  Other Names: PTFE or Cytoplast
  Arms: Non-resorbable membrane
Procedure: Acellular dermal matrix — The ridge preservation graft will be covered with an acellular dermal matrix allograft during the surgery.
  Other Names: Acellular dermal matrix allograft, Alloderm
  Arms: Acellular dermal matrix

SUMMARY:
The purpose of this study is to compare the clinical and histologic outcomes for acellular dermal matrix and a nonresorbable membrane to determine if either provides a significant therapeutic advantage. The hypothesis is that there will be no difference in crestal ridge width between the two treatments.

DETAILED DESCRIPTION:
30 patients will be selected that meet the following criteria:

Inclusion Criteria

1. Have one non-molar tooth requiring extraction that will be replaced by a dental implant. The site must be bordered by at least one tooth.
2. Healthy male or female who is at least 18 years old.
3. Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria

1. Patients with debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium.
2. Presence or history of osteonecrosis of jaws.
3. Patients who are currently taking IV bisphosphonates or who had IV treatment with bisphosphonates irrespective of duration.
4. Patients who have been treated with oral bisphosphonates for more than three years.
5. Patients with an allergy to any material or medication used in the study.
6. Patients who need prophylactic antibiotics.
7. Previous head and neck radiation therapy.
8. Chemotherapy in the previous 12 months.
9. Patients on long term NSAID or steroid therapy.
10. Pregnant patients.

ELIGIBILITY:
Inclusion Criteria:

1. Have one non-molar tooth requiring extraction that will be replaced by a dental implant. The site must be bordered by at least one tooth.
2. Healthy male or female who is at least 18 years old.
3. Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

1. Patients with debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium.
2. Presence or history of osteonecrosis of jaws.
3. Patients who are currently taking IV bisphosphonates or who had IV treatment with bisphosphonates irrespective of duration.
4. Patients who have been treated with oral bisphosphonates for more than three years.
5. Patients with an allergy to any material or medication used in the study.
6. Patients who need prophylactic antibiotics.
7. Previous head and neck radiation therapy.
8. Chemotherapy in the previous 12 months.
9. Patients on long term NSAID or steroid therapy.
10. Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Crestal ridge width | 4 months
  The width of the ridge at the crest will be measured with a digital caliper.

SECONDARY OUTCOMES:
Percent vital bone | 4 months
  Percent vital bone at the graft site will be determined from a trephine core sample.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics Clinic University of Louisville, Louisville, Kentucky, United States